CLINICAL TRIAL: NCT06640582
Title: Efficacy and Safety of Autologous Tumor-Infiltrating Lymphocytes (TIL) Therapy Combined With Pembrolizumab Immunotherapy in Patients With Advanced Brain Cancer Including Gliomas and Meningiomas
Brief Title: TIL Therapy Combined With Pembrolizumab for Advanced Brain Cancer Including Gliomas and Meningiomas
Acronym: BAH2472
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Essen Biotech (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESBI202473
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Brain Tumor; Brain Metastases; Brain Cancer; Glioma; Gliomas, Malignant; Glioblastoma; Meningioma
Keywords: Tumor Infiltrating Lymphocytes; CAR-T CELL; Biological Therapy; Advanced or Metastatic Refractory; Immunotherapy; TIL
MeSH Terms: conditions — Brain Neoplasms; Glioma; Glioblastoma; Meningioma | interventions — Cyclophosphamide; fludarabine; Interleukin-2; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biological Tumor Infiltrating Lymphocytes (TIL) Therapy with Immunotherapy (Experimental): Patients receive pembrolizumab IV on day -14, cyclophosphamide IV QD on days -7 to -6, fludarabine IV over 30 minutes QD on days -5 to -1, and TILs IV infusion on day 0. Patients also receive pembrolizumab IV on day 28 and 70, and undergo surgery on day 80.
  MAINTENANCE: Patients receive pembrolizumab IV every 6 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Tumor Infiltrating Lymphocytes (TIL); Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Interleukin-2; Drug: Pembrolizumab

INTERVENTIONS:
Biological: Tumor Infiltrating Lymphocytes (TIL) — Tumor Infiltrating Lymphocytes (TIL) IV
Drug: Cyclophosphamide — Cyclophosphamide will be administered as an intravenous (IV) infusion for two days.
Drug: Fludarabine — Fludarabine will be administered as an intravenous (IV) infusion for five days.
Drug: Interleukin-2 — After TIL infusion, IL-2 will be started as a bolus administration every eight hours, for a maximum of eight doses.
Drug: Pembrolizumab — Intravenous (IV) infusion

SUMMARY:
This Phase I/II study evaluates the safety and efficacy of autologous tumor-infiltrating lymphocytes (TIL) therapy combined with Pembrolizumab (Keytruda) immunotherapy in patients with Advanced Brain Cancer including Gliomas and Meningiomas . Lifileucel (Amtagvi), the first FDA-approved TIL therapy, has demonstrated significant success in treating unresectable or metastatic melanoma by utilizing the patient's own immune cells to combat cancer. This study aims to apply a similar approach to Brain cancer. TILs will be harvested from patients' tumors, expanded in vitro, and infused back into the patients following a non-myeloablative lymphodepletion regimen. Pembrolizumab, a monoclonal antibody targeting the PD-1 receptor on T cells, will be administered to enhance the immune response. The primary endpoint is to determine the objective response rate (ORR) of this combined therapy. Secondary endpoints include disease control rate (DCR), progression-free survival (PFS), overall survival (OS), duration of response (DOR), and quality of life (QoL). This trial aims to offer a novel, personalized treatment option for patients with limited therapeutic alternatives.

DETAILED DESCRIPTION:
Tumor-infiltrating lymphocytes (TILs) therapy is an innovative form of adoptive cell therapy that utilizes the patient's own immune cells to target and destroy cancer cells. Lifileucel (Amtagvi), the first FDA-approved TIL therapy, has shown remarkable efficacy in treating unresectable or metastatic melanoma. By extracting lymphocytes from the patient's tumor, expanding them ex vivo, and reinfusing them, Lifileucel has significantly improved the immune system's ability to combat cancer cells. This promising approach forms the basis for this study, which aims to apply similar methodologies to advanced or metastatic refractory lung cancer, a condition that generally has a poor prognosis and limited treatment options.

This trial involves several steps: initially, tumor samples are collected from patients for TIL extraction. Afterward, a lymphodepletion regimen using cyclophosphamide and fludarabine is administered to prepare the body for the infusion of expanded autologous TILs. Following the TIL infusion, Aldesleukin (IL-2) is administered to stimulate the TILs' activity. Pembrolizumab (Keytruda), an immunotherapy targeting the PD-1 receptor on T cells, is also given to further enhance the immune response against the tumor.

The primary goal of this trial is to determine the objective response rate (ORR) of this combined therapy. Secondary endpoints include the disease control rate (DCR), progression-free survival (PFS), overall survival (OS), duration of response (DOR), and changes in the quality of life (QoL) of patients.

Patients will be closely monitored for side effects and reactions during their hospital stay and throughout the follow-up period. Safety will be assessed based on the incidence and severity of adverse events, while efficacy will be evaluated using RECIST v1.1 criteria. By leveraging the patient's own immune cells and combining them with advanced immunotherapies, this trial aims to provide a novel, personalized treatment option for patients with advanced or metastatic refractory lung cancer, building on the success observed with Lifileucel (Amtagvi) in melanoma treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age: 16 years to 90 years
* Histologically diagnosed as primary/relapsed/metastasized brain glioma
* Expected life span more than 3 months
* Karnofsky≥60% or ECOG score 0-2
* Test subjects have failed standard treatment regimens, or there are no standard treatment regimens available.
* Test subjects must have tumor regions eligible for biopsy or resection, or malignant body fluid where TILs can be isolated
* At least 1 evaluable tumor lesion
* Hematology and Chemistry（within 7 days prior to enrollment）:
* Absolute count of white blood cells≥2.5×10^9/L
* Absolute count of neutropils≥1.5×10^9/L
* Absolute count of lymphocytes ≥0.7×109/L
* Platelet count≥100×10^9
* hemoglobin≥90 g/L
* Activated partial thromboplastin time (APTT) ≤1.5xULN (Unless received anticoagulant therapy within the previous 3 days)
* International normalized ratio (INR) ≤1.5xULN (Unless received anticoagulant therapy within the previous 3 days)
* Serum creatinine ≤1.5mg/dL(or ≤132.6μmol/L), or clearance rate≥50mL/min
* Serum ALT/AST ≤3×ULN(subjects with liver metastasis ≤3×ULN)
* Totol bilirubin≤1.5×ULN
* No absolute or relative contraindications to operation or biopsy
* Test subjects with child-bearing potential must be willing to practice approved highly effective methods of contraception at the time of informed consent and continue within 1 year after the completion of lymphodepletion
* Any malignant tumor-targeting therapies, including radiotherapy, chemotherapy, and biologics must cease 28 days before obtaining TILs
* Be able to understand and sign the informed consent document;
* Be able to stick to follow-up visit plan and other requirements in the agreement.

Exclusion Criteria:

* Need glucocorticoid treatment, and daily dose of Prednisone greater than 15mg (or equivalent doses of hormones) or outoimmune diseases requiring immunomodulatory treatment
* Forced expiratory volume in one second (FEV1) less than 2L, diffusing capacity of the lung for carbon monoxide (DLCO) (calibrated) less than 40%
* Significant cardiovascular anomalies according to any of the following definitions:
* New York Heart Association (NYHA) Grade III or IV congestive heart failure, clinically significant
* Low blood pressure, uncontrollable symptomatic coronary artery diseases, or ejection fraction less than 35%; Severe cardiac rhythm and conduction anomaly, such as ventricular arrhythmia requiring clinical intervention, second-third degree atrioventricular conductive block, etc.
* Human immunodeficiency virus (HIV) infection or anti-HIV antibody positive, active HBV or HCV infection (HBsAg positive and/or anti-HCV positive), syphilis infection or Treponema pallidum antibody positive.
* Severe physical or mental diseases;
* Have a systemic active infection requiring treatment, or have positive blood cultures(or imaging evidence of infection).
* Having been treated within a month or being treated now with other medicines, or other biologic therapy, chemo-or radiotherapy.
* History of allergy to chemical compounds consisting of chemical and biological substances resembling cell therapy.
* Having received immunotherapy and developed an irAE level greater than Level 3.
* Previous anti-tumor treatment AE did not return to CTCAE5.0 version grade 1 or below (toxicity considered by the investigator as non-safety concerns like alopecia excluded).
* Females in pregnancy or lactation. History of organ transplantation, allogeneic stem cell transplantation, and renal replacement therapy.
* Researchers consider the test subject as having a history of other severe systemic diseases, or other reasons inappropriate for the clinical study.

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2024-10-20 (Actual); Primary Completion 2026-09-10 (Estimated); Study Completion 2026-12-28 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 6 months
  To characterize the safety profile of (TIL) and natural autologous TIL in patients with advanced solid tumors who were failed to standard treatment as assessed by incidence of adverse events.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 36 months
  Proportion of patients with response per Response Evaluation Criteria in Solid Tumors
Disease Control Rate (DCR） | Up to 36 months
  Percentage of patients that meet CR, PR and SD criteria set in this study
Duration of Response (DOR) | Up to 36 months
  The time length between the first confirmed objective response to the treatment and the subsequent disease progression
Progression-Free Survival (PFS) | Up to 36 months
  The time length between TIL infusion and confirmed subsequent disease progression

CONTACTS AND LOCATIONS:
Locations (1):
- District One Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No